CLINICAL TRIAL: NCT07347496
Title: A Randomized, Single-blind, Parallel-controlled Clinical Study to Evaluate the Safety and Efficacy of Remimazolam Besylate Combined With Alfentanil in Anesthesia for Thoracic Surgery
Brief Title: A Randomized, Controlled Clinical Trial Comparing Remimazolam Besylate Combined With Alfentanil Versus Propofol Combined With Alfentanil for Anesthesia in Thoracic Surgery
Acronym: RAA-TS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HNMU-RAA-TS-2026-001
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Thoracic Surgery; Anesthesia; Non-intubated Anesthesia
Keywords: Remimazolam; Alfentanil; Propofol; Non-intubated; Tubeless Anesthesia; Spontaneous Ventilation Spontaneous Ventilation; Total Intravenous Anesthesia Total Intravenous Anesthesia
MeSH Terms: interventions — Injections; Propofol; Alfentanil

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-blind, parallel-group, controlled, superiority trial. Participants will be allocated in a 1:1 ratio to receive either the experimental regimen (Remimazolam Besylate combined with Alfentanil) or the active comparator regimen (Propofol combined with Alfentanil) for anesthesia maintenance during non-intubated video-assisted thoracic surgery.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a single-blind study. Participants (patients) and the research personnel responsible for outcome assessment (e.g., collecting postoperative recovery data, evaluating complications) will be blinded to group assignment.
  The anesthesiologists administering the anesthetic drugs cannot be blinded due to the clinical requirements for drug titration and patient safety management.
  To minimize potential bias, all syringes and infusion lines will be covered with opaque labels to conceal the study drug's appearance from the participant and assessment staff. Standardized anesthesia and surgical protocols will be strictly followed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam Besylate + Alfentanil (Experimental): Patients will receive total intravenous anesthesia induced and maintained with Remimazolam Besylate in combination with Alfentanil.
  Interventions: Drug: Propofol; Drug: Alfentanil Hydrochloride Injection
- Propofol + Alfentanil (Active Comparator): Patients will receive total intravenous anesthesia induced and maintained with Propofol in combination with Alfentanil (standard care).
  Interventions: Drug: Remimazolam Besylate for Injection; Drug: Alfentanil Hydrochloride Injection

INTERVENTIONS:
Drug: Remimazolam Besylate for Injection — A novel ultra-short-acting benzodiazepine. Induction dose: 0.3 mg/kg. Maintenance: continuous infusion at 0.2-1 mg/kg/h, titrated to maintain a BIS value between 40-60.
  Arms: Propofol + Alfentanil
Drug: Propofol — Standard intravenous anesthetic. Induction dose: 1.5-2 mg/kg. Maintenance: continuous infusion at 2-6 mg/kg/h, titrated to maintain a BIS value between 40-60.
  Arms: Remimazolam Besylate + Alfentanil
Drug: Alfentanil Hydrochloride Injection — A short-acting opioid analgesic. Administered at induction (10 μg/kg) and as a continuous infusion (0-1 μg/kg/min) for intraoperative analgesia.

SUMMARY:
Title: A Clinical Study Comparing Two Anesthesia Methods for Chest Surgery

Why is this study being done? Chest surgeries (like lung surgery) require safe and stable anesthesia. Currently, a drug called propofol combined with an opioid painkiller (alfentanil) is commonly used. However, propofol can sometimes cause low blood pressure and low oxygen levels. A newer drug called remimazolam may cause fewer of these side effects. This study aims to compare the safety and effectiveness of remimazolam (combined with alfentanil) versus propofol (combined with alfentanil) for anesthesia during chest surgery.

What will happen in the study?

Patients scheduled for elective chest surgery will be invited to participate. If they agree, they will be randomly assigned (like flipping a coin) to one of two groups:

* Group 1: Will receive remimazolam and alfentanil for anesthesia.
* Group 2: Will receive propofol and alfentanil for anesthesia (standard care).

The anesthesiologist will carefully monitor patients during and after surgery. We will mainly compare how often patients in each group experience two safety issues: low oxygen levels in the blood and low blood pressure. We will also record recovery times, drug doses, side effects, and ask patients and surgeons about their satisfaction.

Who can participate? Adults aged 18-65 who are scheduled for elective chest surgery and are in relatively stable health (ASA physical status I-III).

Where is the study taking place? This study will be conducted in the Department of Anesthesiology at The First Affiliated Hospital of Xinxiang Medical College, Henan, China.

Ethics Approval:

This study has been reviewed and approved by the Ethics Committee of The First Affiliated Hospital of Xinxiang Medical College (Approval Number: (2025) Medical Ethics Committee Approval No. 29).

DETAILED DESCRIPTION:
Study Design:

This is a prospective, randomized, single-blind, parallel-group, controlled clinical trial. It is designed as a Phase IV study comparing the clinical profiles of two established anesthetic regimens.

Background and Rationale:

Thoracic surgery, particularly procedures requiring one-lung ventilation, poses significant challenges for anesthetic management, demanding excellent hemodynamic stability and respiratory control. Propofol, while a mainstay for total intravenous anesthesia, is associated with dose-dependent hypotension and respiratory depression. Remimazolam, a novel ultrashort-acting benzodiazepine, is metabolized by tissue esterases and may offer a more stable hemodynamic profile. Combining it with the short-acting opioid alfentanil could provide an effective and potentially safer alternative for thoracic anesthesia. This study seeks to generate high-level evidence comparing these two combinations in a surgical setting known for its physiological demands.

Intervention Protocol:

* Premedication & Induction: All patients will receive standardized premedication. Anesthesia induction will begin with alfentanil (10 μg/kg), followed by the study drug: either Remimazolam Besylate (0.3 mg/kg) or Propofol (1.5-2 mg/kg).
* Maintenance: Anesthesia will be maintained via continuous infusion of the assigned study drug (Remimazolam: 0.2-1 mg/kg/h; Propofol: 2-6 mg/kg/h) along with alfentanil (0-1 μg/kg/min), titrated to maintain a Bispectral Index (BIS) value between 40-60.
* Standardization: All patients will undergo standardized monitoring, airway management, and surgical and analgesic protocols as per institutional guidelines for thoracic surgery.

Primary Objectives:

To compare the incidence of intraoperative hypoxemia (SpO₂ < 90% for >10 seconds) and intraoperative hypotension (MAP < 65 mmHg or a decrease >20% from baseline) between the two groups.

Key Secondary Objectives:

Include comparison of: hemodynamic variables, need for rescue interventions, times to extubation and recovery, total drug consumption, incidence of postoperative nausea/vomiting (PONV), postoperative pulmonary complications, quality of recovery (QoR-15), and satisfaction scores from patients and surgeons.

Statistical Analysis:

Data will be analyzed based on the Intention-to-Treat principle. Categorical data will be compared using Chi-square or Fisher's exact test. Continuous data will be analyzed using Student's t-test or Mann-Whitney U test, as appropriate. Subgroup analyses are planned for specific patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective thoracic surgery (e.g., pulmonary lobectomy, esophagectomy) under general anesthesia with preserved spontaneous respiration.
* American Society of Anesthesiologists (ASA) physical status class I-III.
* Age between 18 and 75 years.
* Provide written informed consent.

Exclusion Criteria:

* Severe hepatic or renal dysfunction (e.g., Child-Pugh class C, eGFR < 30 mL/min/1.73m²).
* Severe respiratory dysfunction (e.g., COPD GOLD stage 3-4, severe asthma).
* Anticipated difficult airway (e.g., Mallampati class IV, history of difficult intubation).
* Known allergy or hypersensitivity to benzodiazepines, opioids, or propofol.
* Pregnancy or lactation.
* Participation in another interventional clinical trial within the past 3 months.
* Mental illness or inability to cooperate with assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Intraoperative Hypoxemia | From induction of anesthesia until the end of surgery.
  Defined as peripheral oxygen saturation (SpO₂) < 90% for more than 10 seconds during surgery.
Incidence of Intraoperative Hypotension | From induction of anesthesia until the end of surgery.
  Defined as mean arterial pressure (MAP) < 65 mmHg or a decrease >20% from baseline during surgery.

SECONDARY OUTCOMES:
Need for Airway Maneuver | From induction of anesthesia until the end of surgery.
Time to Extubation | From induction of anesthesia until the end of surgery.
Incidence of Postoperative Nausea and Vomiting (PONV) | From induction of anesthesia until the end of surgery.
Patient Satisfaction Score | From induction of anesthesia until the end of surgery.